CLINICAL TRIAL: NCT01174069
Title: Clinical Outcomes Trial of Laparoscopic Assisted Transgastric Endoscopic Cholecystectomy
Brief Title: Natural Orifice Transgastric Endoscopic Surgical Removal of the Gallbladder
Acronym: NOTESchole
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Oregon Clinic (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Lee Swanstrom, MD, The Oregon Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LHS0701
Record Dates: First submitted 2010-07-30; First posted 2010-08-03 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Cholecystitis
Keywords: NOTES; cholecystectomy; endoscopic
MeSH Terms: conditions — Cholecystitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NOTES cholecystectomy (Experimental)
  Interventions: Procedure: NOTES assisted laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: NOTES assisted laparoscopic cholecystectomy — Surgical removal of the gallbladder using endoscopic instruments.
  Other Names: NOTES Cholecystectomy

SUMMARY:
Hypothesis: Natural orifice transgastric cholecystectomy with laparoscopic assist will be feasible and have comparable complication rates as standard lap cholecystectomy. Patient benefits will include less pain and scaring.

DETAILED DESCRIPTION:
In this study, we propose to use a surgical technique that eliminates the need for a 1.5-2.5 cm umbilical incision. A flexible endoscope will be inserted through the mouth and into the stomach. Using commercially available endoscopes, endoscopic instruments and accessories, a small incision will be made in the gastric wall and the endoscope will be advanced into the insufflated peritoneal cavity. Two to three small laparoscopic trocars will be placed for laparoscopic instrument insertion to manipulate, retract and cut tissue. The flexible endoscope will provide visualization of the surgical field and flexible endoscopic instruments may be used to augment surgical manipulation with the laparoscopic instruments. Once dissected free, the gall bladder will be removed through the stomach and out of the mouth. Commercially available endoscopic clips, sutures and/or tissue anchors will be used to close the gastrotomy; additionally, the gastrotomy will be tested for leaks and laparoscopically oversewn with suture as needed.

Patients will be discharged per the standard of practice for a laparoscopic cholecystectomy. During the hospital stay severity of pain and use of pain medications will be recorded. Length of time spent in the recovery room and in the hospital will also be collected. Patients will return and be evaluated by their surgeon two weeks following their procedure. At this visit, any complications will be noted in the patient's medical record. Additionally at this visit and at the preoperative visit, patients will complete a standardized Quality of Life (QOL) assessment (i.e., SF-36) and perceived pain levels and type and frequency of pain medications will be recorded in the patient's medical record.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to undergo general anesthesia
2. Age > 18 years of age and < 80 years of age
3. Ability to give informed consent

Exclusion Criteria:

1. Acute cholecystitis
2. Body Mass Index (BMI) > 40
3. Contraindicated for esophagogastroduodenoscopy (EGD)
4. Gallstones > 2.5cm in diameter
5. Gall bladder more than 15cm in length on U/S
6. Presence of common duct stones
7. Presence of esophageal stricture
8. Altered gastric anatomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 30 days
  perceived pain levels and type and frequency of pain medications will be recorded in the patient's medical record.

SECONDARY OUTCOMES:
Perception of surgical outcome | 30 days post operatively
  standardized Quality of Life (QOL) assessment (i.e., SF-36) form filled out by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Christy M Dunst, MD, Principal Investigator — The Oregon Clinic; Angi B Gill, RN, Study Director — The Oregon Clinic
Locations (1):
- Legacy health System, Portland, Oregon, United States